CLINICAL TRIAL: NCT00211016
Title: A Multicenter, Randomized, Open-Label, Phase 3 Study of Doripenem Versus a Comparator Antibiotic in the Treatment of Ventilator-Associated Pneumonia
Brief Title: Doripenem in the Treatment of Ventilator-Associated Pneumonia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Collaborators: Peninsula Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005386
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2010-03

CONDITIONS: Pneumonia; Ventilators, Mechanical
Keywords: Ventilator-Associated Pneumonia
MeSH Terms: conditions — Pneumonia; Pneumonia, Ventilator-Associated | interventions — Doripenem

INTERVENTIONS:
Drug: doripenem

SUMMARY:
The purpose of this study is to compare the clinical response rate of doripenem versus comparator in patients with ventilator-associated pneumonia (VAP).

DETAILED DESCRIPTION:
Doripenem is an antibiotic medication not yet approved by the US FDA. This is a phase 3, multicenter, prospective, randomized, open-label study of doripenem versus comparator to assess the effectiveness and safety of doripenem in the treatment of VAP in adult patients. The study consists of screening phase, open-label treatment phase, and follow-up. The treatment duration is from 7 to 14 days. The primary endpoint is the clinical response rate of doripenem at the early follow-up visit. The patients will receive either doripenem or comparator for 7 to 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient has received mechanical ventilation for > 24 hours
* Presence of a new or progressive infiltrate on chest x-ray

Exclusion Criteria:

* Believed at study entry to have ventilator-associated pneumonia caused solely by pathogen(s) resistant to certain antibiotics
* History of moderate or severe hypersensitivity reactions to certain antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2004-08; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Clinical response rate at the early follow-up visit.

SECONDARY OUTCOMES:
Clinical response rate at the late follow-up visit. Microbiological response at both early and late follow-up visits. Safety assessment (adverse events, vital signs, laboratory test results) conducted throughout the study..

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Kollef MH, Nathwani D, Merchant S, Gast C, Quintana A, Ketter N. Medical resource utilization among patients with ventilator-associated pneumonia: pooled analysis of randomized studies of doripenem versus comparators. Crit Care. 2010;14(3):R84. doi: 10.1186/cc9012. Epub 2010 May 10. PMID 20459721
- [Derived] Kaniga K, Flamm R, Tong SY, Lee M, Friedland I, Redman R. Worldwide experience with the use of doripenem against extended-spectrum-beta-lactamase-producing and ciprofloxacin-resistant Enterobacteriaceae: analysis of six phase 3 clinical studies. Antimicrob Agents Chemother. 2010 May;54(5):2119-24. doi: 10.1128/AAC.01450-09. Epub 2010 Mar 8. PMID 20211892
- [Derived] Zhanel GG, Ketter N, Rubinstein E, Friedland I, Redman R. Overview of seizure-inducing potential of doripenem. Drug Saf. 2009;32(9):709-16. doi: 10.2165/00002018-200932090-00001. PMID 19670912
- See also: A Multicenter, Randomized, Open-Label, Phase 3 Study to Compare the Safety and Efficacy of Intravenous Doripenem with that of Intravenous Imipenem in Ventilator-Associated Pneumonia — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=638&filename=CR005386_CSR.pdf